CLINICAL TRIAL: NCT02481193
Title: Effects of Cisatracurium on Succinylcholine-induced Fasciculations and Myalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yangzhou No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Dongsheng Zhang, MD, MD, Yangzhou No.1 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YZYY-610
Record Dates: First submitted 2015-06-10; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Fasciculation
Keywords: Cisatracurium; Myalgia; Fasciculation; Succinylcholine
MeSH Terms: conditions — Fasciculation; Myalgia | interventions — cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cisatracurium 0.005 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.005 mg/kg.
  Interventions: Drug: Cisatracurium
- Cisatracurium 0.01 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.01 mg/kg
  Interventions: Drug: Cisatracurium
- Cisatracurium 0.02 mg/kg (Experimental): The group received pretreatment of cisatracurium 0.02 mg/kg
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — Different doses of cisatracurium pretreatment
  Other Names: Dose

SUMMARY:
The purpose of this study is to investigate the effects of different doses of cisatracurium pretreatment on succinylcholine-induced fasciculations and postoperative myalgia.

DETAILED DESCRIPTION:
Purpose: To investigate the effects of different doses of cisatracurium pretreatment on succinylcholine-induced fasciculations and postoperative myalgia.

Methods: Ninety patients scheduled for laparoscopic cholecystectomies were equally randomized into three groups to receive pretreatment of 0.005, 0.01, and 0.02 mg/kg cisatracurium, respectively. General anesthesia was induced 3.5 min later, train of four stimulation was monitored 4.5 min later, succinylcholine 1.5 mg/kg was injected 5 min later, and endotracheal intubation was implemented 6.5 min later. The side effects of cisatracurium, intensity of fasciculations, intubating conditions, time and extent to maximal depression of twitch and time for its recovery to 20% of control value, severity of myalgia at 24 h postoperatively, serum potassium before the induction, at the time of endotracheal intubation, and 5 min after intubation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Standards Association (ASA) physical status I or II patients scheduled for elective laparoscopic cholecystectomies with tracheal intubation requiring general anesthesia
* 20 - 65 years old
* without acid-base imbalance and electrolyte disturbance
* with normal hepatic and renal function

Exclusion Criteria:

* Patients with known hyperkalemia
* Patients with increased intraocular pressure
* Patients with increased intracranial pressure
* Patients with symptoms of gastroesophageal reflux
* Patients with anticipated airway difficulties
* Patients with malignant fever
* Patients with neuromuscular disease
* Patients with burn or crush injuries
* Patients with taking drugs known to alter the action of neuromuscular blockers
* Patients with with a body mass index exceeding 30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The presence of fasciculations | After the injection of succinylcholine for 1.5 minutes

SECONDARY OUTCOMES:
Side effects of the pretreatment of cisatracurium | At the time of three minutes after the pretreatment of cisatracurium
The time to maximal depression of twitch | From the time of 4.5 minutes after the pretreatment of cisatracurium for two minutes
The extent to maximal depression of twitch | From the time of 4.5 minutes after the pretreatment of cisatracurium for two minutes
The time for twitch recovery to 20% of its control value | From the time of 4.5 minutes after the pretreatment of cisatracurium for two minutes
The grades of endotracheal intubation | At intubating time
The changes of serum potassium | After entering the operating theater till the anesthesia induction, at intubating, and 5 min after intubation
Myalgia at 24 hours postoperatively | At 24 hours postoperatively